CLINICAL TRIAL: NCT01865617
Title: Phase I/II Study of Immunotherapy for Advanced CD19+ Chronic Lymphocytic Leukemia, Acute Lymphoblastic Leukemia/Lymphoma and Non-Hodgkin Lymphoma With Defined Subsets of Autologous T Cells Engineered to Express a CD19-Specific Chimeric Antigen Receptor
Brief Title: Laboratory Treated T Cells in Treating Patients With Relapsed or Refractory Chronic Lymphocytic Leukemia, Non-Hodgkin Lymphoma, or Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Alexandre Hirayama, Research Associate, Fred Hutchinson Cancer Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2639.00; NCI-2013-00073 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2639; RG9213011 (Other: Fred Hutch/University of Washington Cancer Consortium); P50CA107399 (NIH); R01CA136551 (NIH)
Record Dates: First submitted 2013-05-28; First posted 2013-05-31 (Estimated); Results first posted 2022-05-25 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: CD19-Positive Neoplastic Cells Present; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Chronic Lymphocytic Leukemia; Recurrent Diffuse Large B-Cell Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Non-Hodgkin Lymphoma; Recurrent Small Lymphocytic Lymphoma; Refractory Acute Lymphoblastic Leukemia; Refractory Chronic Lymphocytic Leukemia; Refractory Diffuse Large B-Cell Lymphoma; Refractory Mantle Cell Lymphoma; Refractory Non-Hodgkin Lymphoma; Refractory Small Lymphocytic Lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (13):
- ALL (high tumor burden) dose level 1 (Experimental): Patients receive anti-CD19-CAR lentiviral vector-transduced autologous T cells IV over 20-30 minutes on day 0. Treatment may be repeated in no less than 21 days with or without additional lymphodepleting chemotherapy if there is persistent disease in the absence of unacceptable toxicity.
  Disease subgroup: ALL Tumor Burden: high Dose level: 1 up to 2x105 EGFR+ cells/kg
  Interventions: Biological: Autologous Anti-CD19CAR-4-1BB-CD3zeta-EGFRt-expressing T Lymphocytes
- ALL (high tumor burden) dose level 2 (Experimental): Patients receive anti-CD19-CAR lentiviral vector-transduced autologous T cells IV over 20-30 minutes on day 0. Treatment may be repeated in no less than 21 days with or without additional lymphodepleting chemotherapy if there is persistent disease in the absence of unacceptable toxicity.
  Disease subgroup: ALL Tumor Burden: high Dose level: 2 up to 2x106 EGFR+ cells/kg
  Interventions: Biological: Autologous Anti-CD19CAR-4-1BB-CD3zeta-EGFRt-expressing T Lymphocytes
- ALL (high tumor burden) dose level 3 (Experimental): Patients receive anti-CD19-CAR lentiviral vector-transduced autologous T cells IV over 20-30 minutes on day 0. Treatment may be repeated in no less than 21 days with or without additional lymphodepleting chemotherapy if there is persistent disease in the absence of unacceptable toxicity.
  Disease subgroup: ALL Tumor Burden: high Dose level: 3 up to 2x107 EGFR+ cells/kg
  Interventions: Biological: Autologous Anti-CD19CAR-4-1BB-CD3zeta-EGFRt-expressing T Lymphocytes
- ALL (low tumor burden) dose level 1 (Experimental): Patients receive anti-CD19-CAR lentiviral vector-transduced autologous T cells IV over 20-30 minutes on day 0. Treatment may be repeated in no less than 21 days with or without additional lymphodepleting chemotherapy if there is persistent disease in the absence of unacceptable toxicity.
  Disease subgroup: ALL Tumor Burden: low Dose level: 1 up to 2x105 EGFR+ cells/kg
  Interventions: Biological: Autologous Anti-CD19CAR-4-1BB-CD3zeta-EGFRt-expressing T Lymphocytes
- ALL (low tumor burden) dose level 2 (Experimental): Patients receive anti-CD19-CAR lentiviral vector-transduced autologous T cells IV over 20-30 minutes on day 0. Treatment may be repeated in no less than 21 days with or without additional lymphodepleting chemotherapy if there is persistent disease in the absence of unacceptable toxicity.
  Disease subgroup: ALL Tumor Burden: high Dose level: 2 up to 2x106 EGFR+ cells/kg
  Interventions: Biological: Autologous Anti-CD19CAR-4-1BB-CD3zeta-EGFRt-expressing T Lymphocytes
- CLL dose level 1 (Experimental): Patients receive anti-CD19-CAR lentiviral vector-transduced autologous T cells IV over 20-30 minutes on day 0. Treatment may be repeated in no less than 21 days with or without additional lymphodepleting chemotherapy if there is persistent disease in the absence of unacceptable toxicity.
  Disease subgroup: CLL Dose level: 1 up to 2x105 EGFR+ cells/kg
  Interventions: Biological: Autologous Anti-CD19CAR-4-1BB-CD3zeta-EGFRt-expressing T Lymphocytes
- CLL dose level 2 (Experimental): Patients receive anti-CD19-CAR lentiviral vector-transduced autologous T cells IV over 20-30 minutes on day 0. Treatment may be repeated in no less than 21 days with or without additional lymphodepleting chemotherapy if there is persistent disease in the absence of unacceptable toxicity.
  Disease subgroup: CLL Dose level: 2 up to 2x106 EGFR+ cells/kg
  Interventions: Biological: Autologous Anti-CD19CAR-4-1BB-CD3zeta-EGFRt-expressing T Lymphocytes
- CLL dose level 3 (Experimental): Patients receive anti-CD19-CAR lentiviral vector-transduced autologous T cells IV over 20-30 minutes on day 0. Treatment may be repeated in no less than 21 days with or without additional lymphodepleting chemotherapy if there is persistent disease in the absence of unacceptable toxicity.
  Disease subgroup: CLL Dose level: 3 up to 2x107 EGFR+ cells/kg
  Interventions: Biological: Autologous Anti-CD19CAR-4-1BB-CD3zeta-EGFRt-expressing T Lymphocytes
- CLL (ibrutinib) dose level 2 (Experimental): Patients receive anti-CD19-CAR lentiviral vector-transduced autologous T cells IV over 20-30 minutes on day 0. Treatment may be repeated in no less than 21 days with or without additional lymphodepleting chemotherapy if there is persistent disease in the absence of unacceptable toxicity.
  Disease subgroup: CLL (ibrutinib) Dose level: 2 up to 2x106 EGFR+ cells/kg
  Interventions: Biological: Autologous Anti-CD19CAR-4-1BB-CD3zeta-EGFRt-expressing T Lymphocytes
- NHL dose level 1 (Experimental): Patients receive anti-CD19-CAR lentiviral vector-transduced autologous T cells IV over 20-30 minutes on day 0. Treatment may be repeated in no less than 21 days with or without additional lymphodepleting chemotherapy if there is persistent disease in the absence of unacceptable toxicity.
  Disease subgroup: NHL Dose level: 1 up to 2x105 EGFR+ cells/kg
  Interventions: Biological: Autologous Anti-CD19CAR-4-1BB-CD3zeta-EGFRt-expressing T Lymphocytes
- NHL dose level 2 (Experimental): Patients receive anti-CD19-CAR lentiviral vector-transduced autologous T cells IV over 20-30 minutes on day 0. Treatment may be repeated in no less than 21 days with or without additional lymphodepleting chemotherapy if there is persistent disease in the absence of unacceptable toxicity.
  Disease subgroup: NHL Dose level: 2 up to 2x106 EGFR+ cells/kg
  Interventions: Biological: Autologous Anti-CD19CAR-4-1BB-CD3zeta-EGFRt-expressing T Lymphocytes
- NHL dose level 3 (Experimental): Patients receive anti-CD19-CAR lentiviral vector-transduced autologous T cells IV over 20-30 minutes on day 0. Treatment may be repeated in no less than 21 days with or without additional lymphodepleting chemotherapy if there is persistent disease in the absence of unacceptable toxicity.
  Disease subgroup: NHL Dose level: 3 up to 2x107 EGFR+ cells/kg
  Interventions: Biological: Autologous Anti-CD19CAR-4-1BB-CD3zeta-EGFRt-expressing T Lymphocytes
- NHL (dose dense) dose level 2 (Experimental): Patients receive anti-CD19-CAR lentiviral vector-transduced autologous T cells IV over 20-30 minutes on day 0. Treatment may be repeated in no less than 21 days with or without additional lymphodepleting chemotherapy if there is persistent disease in the absence of unacceptable toxicity.
  Disease subgroup: NHL Dose level: 2 up to 2x106 EGFR+ cells/kg
  Interventions: Biological: Autologous Anti-CD19CAR-4-1BB-CD3zeta-EGFRt-expressing T Lymphocytes

INTERVENTIONS:
Biological: Autologous Anti-CD19CAR-4-1BB-CD3zeta-EGFRt-expressing T Lymphocytes — Given IV

SUMMARY:
This phase I/II trial studies the side effects and best dose of laboratory treated T cells to see how well they work in treating patients with chronic lymphocytic leukemia, non-Hodgkin lymphoma, or acute lymphoblastic leukemia that have come back or have not responded to treatment. T cells that are treated in the laboratory before being given back to the patient may make the body build an immune response to kill cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the feasibility and safety of adoptive T cell therapy using ex vivo expanded autologous CD8 positive (+) and CD4+ CD19 chimeric antigen receptor (CAR)-T cells for patients with advanced CD19+ B cell malignancies.

SECONDARY OBJECTIVES:

I. To determine the duration of in vivo persistence of adoptively transferred T cells, and the phenotype of persisting T cells.

II. To determine if adoptively transferred T cells traffic to the bone marrow and function in vivo.

III. To determine if the adoptive transfer of CD19 CAR-T cells results in depletion of CD19+ B cells in vivo as a surrogate for functional activity.

IV. To determine if the adoptive transfer of CD19 CAR-T cells has antitumor activity in patients with measurable tumor burden prior to T cell transfer.

V. To determine if the adoptive transfer of CD19 CAR-T cells is associated with tumor lysis syndrome.

OUTLINE: This is a phase I, dose-escalation study of autologous CD19 CAR T-cells followed by a phase II study.

Patients receive anti-CD19-CAR lentiviral vector-transduced autologous T cells intravenously (IV) over 20-30 minutes on day 0. Treatment may be repeated in no less than 21 days with or without additional lymphodepleting chemotherapy if there is persistent disease in the absence of unacceptable toxicity.

DOSE DENSE EXPANSION COHORT: An additional cohort will receive a second anti-CD19-CAR lentiviral vector-transduced autologous T cell infusion without additional lymphodepleting chemotherapy 10-21 days after the first infusion if adequate CD19 CAR-T cells can be produced and appropriate criteria are met.

After completion of study treatment, patients are followed up for at least 15 years.

ELIGIBILITY:
Inclusion Criteria:

INCLUSIONS FOR SCREENING AND LEUKAPHERESIS

* Patients with CD19 expressing acute lymphoblastic leukemia (ALL), chronic lymphocytic leukemia (CLL) or non-Hodgkin lymphoma (NHL)
* Ability to understand and provide informed consent
* Not human immunodeficiency virus (HIV) infected

INCLUSIONS FOR CAR-T CELL THERAPY

* Patients with:

  * CLL who are beyond first remission and who have failed combination chemoimmunotherapy with regimens containing a purine analogue and anti-CD20 antibody or who were not eligible for such therapy; patients with CLL for whom ibrutinib is now standard first line therapy, must have progressed on ibrutinib; patients with fludarabine refractory disease are eligible; patients may be treated following allogeneic hematopoietic cell transplant (HCT); for the concurrent ibrutinib cohort, patients must agree to continue on or be restarted on ibrutinib and must not have had prior intolerance to ibrutinib that would prevent this; patients managed with prior dose reductions for toxicity will continue at the reduced dose for the remainder of this study
  * Indolent NHL or mantle cell NHL who are beyond first remission and previously treated with chemoimmunotherapy or who were not eligible for such therapy; patients who have relapsed following autologous or allogeneic HCT are eligible
  * Aggressive NHL such as diffuse large B-cell lymphoma (DLBCL), who have relapsed or have residual disease following treatment with curative intent; patients should have relapsed following, or not be eligible for high-dose therapy and autologous HCT; patients with chemotherapy refractory disease or marrow involvement or comorbidities precluding successful autologous HCT are eligible; patients may be treated following allogeneic HCT
  * Patients with CD19 expressing, relapsed or refractory ALL
  * Patients with one of the above diagnoses whose disease state does not qualify but who have prognostic indicators that suggest a high risk of progression of disease may be screened and undergo leukapheresis; enrollment for T cell therapy would require meeting the full disease state eligibility
* Confirmation of diagnosis
* Evidence of CD19 expression by immunohistochemistry or flow cytometry on any prior or current tumor specimen or high likelihood of CD19 expression based on disease histology
* Karnofsky performance status >= 60%
* All patients of childbearing potential must be willing to use a contraceptive method before, during, and for at least two months after the T cell infusion
* Ability to understand and provide informed consent

Exclusion Criteria:

EXCLUSIONS FOR CAR-T CELL THERAPY

* Patients requiring ongoing daily corticosteroid therapy at a dose of > 15 mg of prednisone per day (or equivalent); pulsed corticosteroid use for disease control is acceptable
* Active autoimmune disease requiring immunosuppressive therapy is excluded unless discussed with the Principal Investigator (PI)
* Serum creatinine > 2.5 mg/dL
* Serum glutamic oxaloacetic transaminase (SGOT) > 5 x upper limit of normal
* Bilirubin > 3.0 mg/dL
* Patients with clinically significant pulmonary dysfunction, as determined by medical history and physical exam should undergo pulmonary function testing; those with a forced expiratory volume in one second (FEV1) of < 50 % of predicted will be excluded
* Diffusing capacity of the lung for carbon monoxide (DLCO) (corrected) < 40% will be excluded
* Significant cardiovascular abnormalities as defined by any one of the following: New York Heart Association (NYHA) class III or IV congestive heart failure, clinically significant hypotension, uncontrolled symptomatic coronary artery disease, or a documented ejection fraction of < 35%
* Uncontrolled active infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2013-05-22 (Actual); Primary Completion 2021-03-26 (Actual); Study Completion 2021-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Gauthier, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fiorenza S, Zheng Y, Purushe J, Bock TJ, Sarthy J, Janssens DH, Sheih AS, Kimble EL, Kirchmeier D, Phi TD, Gauthier J, Hirayama AV, Riddell SR, Wu Q, Gottardo R, Maloney DG, Yang JYH, Henikoff S, Turtle CJ. Histone marks identify novel transcription factors that parse CAR-T subset-of-origin, clinical potential and expansion. Nat Commun. 2024 Sep 27;15(1):8309. doi: 10.1038/s41467-024-52503-2. PMID 39333103
- [Derived] Liang EC, Albittar A, Huang JJ, Hirayama AV, Kimble EL, Portuguese AJ, Chapuis A, Shadman M, Till BG, Cassaday RD, Milano F, Kiem HP, Riddell SR, Turtle CJ, Maloney DG, Gauthier J. Factors associated with long-term outcomes of CD19 CAR T-cell therapy for relapsed/refractory CLL. Blood Adv. 2023 Nov 28;7(22):6990-7005. doi: 10.1182/bloodadvances.2023011399. PMID 37774014
- [Derived] Juluri KR, Wu QV, Voutsinas J, Hou J, Hirayama AV, Mullane E, Miles N, Maloney DG, Turtle CJ, Bar M, Gauthier J. Severe cytokine release syndrome is associated with hematologic toxicity following CD19 CAR T-cell therapy. Blood Adv. 2022 Apr 12;6(7):2055-2068. doi: 10.1182/bloodadvances.2020004142. PMID 34666344
- [Derived] Ernst M, Oeser A, Besiroglu B, Caro-Valenzuela J, Abd El Aziz M, Monsef I, Borchmann P, Estcourt LJ, Skoetz N, Goldkuhle M. Chimeric antigen receptor (CAR) T-cell therapy for people with relapsed or refractory diffuse large B-cell lymphoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD013365. doi: 10.1002/14651858.CD013365.pub2. PMID 34515338
- [Derived] Gauthier J, Bezerra ED, Hirayama AV, Fiorenza S, Sheih A, Chou CK, Kimble EL, Pender BS, Hawkins RM, Vakil A, Phi TD, Steinmetz RN, Jamieson AW, Bar M, Cassaday RD, Chapuis AG, Cowan AJ, Green DJ, Kiem HP, Milano F, Shadman M, Till BG, Riddell SR, Maloney DG, Turtle CJ. Factors associated with outcomes after a second CD19-targeted CAR T-cell infusion for refractory B-cell malignancies. Blood. 2021 Jan 21;137(3):323-335. doi: 10.1182/blood.2020006770. PMID 32967009
- [Derived] Hirayama AV, Gauthier J, Hay KA, Voutsinas JM, Wu Q, Pender BS, Hawkins RM, Vakil A, Steinmetz RN, Riddell SR, Maloney DG, Turtle CJ. High rate of durable complete remission in follicular lymphoma after CD19 CAR-T cell immunotherapy. Blood. 2019 Aug 15;134(7):636-640. doi: 10.1182/blood.2019000905. PMID 31648294
- [Derived] Hirayama AV, Gauthier J, Hay KA, Voutsinas JM, Wu Q, Gooley T, Li D, Cherian S, Chen X, Pender BS, Hawkins RM, Vakil A, Steinmetz RN, Acharya UH, Cassaday RD, Chapuis AG, Dhawale TM, Hendrie PC, Kiem HP, Lynch RC, Ramos J, Shadman M, Till BG, Riddell SR, Maloney DG, Turtle CJ. The response to lymphodepletion impacts PFS in patients with aggressive non-Hodgkin lymphoma treated with CD19 CAR T cells. Blood. 2019 Apr 25;133(17):1876-1887. doi: 10.1182/blood-2018-11-887067. Epub 2019 Feb 19. PMID 30782611
- [Derived] Tuazon SA, Li A, Gooley T, Eunson TW, Maloney DG, Turtle CJ, Linenberger ML, Connelly-Smith LS. Factors affecting lymphocyte collection efficiency for the manufacture of chimeric antigen receptor T cells in adults with B-cell malignancies. Transfusion. 2019 May;59(5):1773-1780. doi: 10.1111/trf.15178. Epub 2019 Feb 6. PMID 30729531
- [Derived] Hay KA, Gauthier J, Hirayama AV, Voutsinas JM, Wu Q, Li D, Gooley TA, Cherian S, Chen X, Pender BS, Hawkins RM, Vakil A, Steinmetz RN, Schoch G, Chapuis AG, Till BG, Kiem HP, Ramos JD, Shadman M, Cassaday RD, Acharya UH, Riddell SR, Maloney DG, Turtle CJ. Factors associated with durable EFS in adult B-cell ALL patients achieving MRD-negative CR after CD19 CAR T-cell therapy. Blood. 2019 Apr 11;133(15):1652-1663. doi: 10.1182/blood-2018-11-883710. Epub 2019 Feb 6. PMID 30728140
- [Derived] Hill JA, Li D, Hay KA, Green ML, Cherian S, Chen X, Riddell SR, Maloney DG, Boeckh M, Turtle CJ. Infectious complications of CD19-targeted chimeric antigen receptor-modified T-cell immunotherapy. Blood. 2018 Jan 4;131(1):121-130. doi: 10.1182/blood-2017-07-793760. Epub 2017 Oct 16. PMID 29038338
- [Derived] Turtle CJ, Hanafi LA, Berger C, Gooley TA, Cherian S, Hudecek M, Sommermeyer D, Melville K, Pender B, Budiarto TM, Robinson E, Steevens NN, Chaney C, Soma L, Chen X, Yeung C, Wood B, Li D, Cao J, Heimfeld S, Jensen MC, Riddell SR, Maloney DG. CD19 CAR-T cells of defined CD4+:CD8+ composition in adult B cell ALL patients. J Clin Invest. 2016 Jun 1;126(6):2123-38. doi: 10.1172/JCI85309. Epub 2016 Apr 25. PMID 27111235

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 204 patients were enrolled on this study but only 197 met eligibility criteria and went on to be treated on study.
Groups:
- ALL (High Tumor Burden) Dose Level 1: Patients receive anti-CD19-CAR lentiviral vector-transduced autologous T cells IV over 20-30 minutes on day 0. Treatment may be repeated in no less than 21 days with or without additional lymphodepleting chemotherapy if there is persistent disease in the absence of unacceptable toxicity.
  Disease subgroup: ALL Tumor Burden: high Dose level: 1 up to 2x105 EGFR+ cells/kg
  Autologous Anti-CD19CAR-4-1BB-CD3zeta-EGFRt-expressing T Lymphocytes: Given IV
- ALL (High Tumor Burden) Dose Level 2; ALL (Low Tumor Burden) Dose Level 2: Patients receive anti-CD19-CAR lentiviral vector-transduced autologous T cells IV over 20-30 minutes on day 0. Treatment may be repeated in no less than 21 days with or without additional lymphodepleting chemotherapy if there is persistent disease in the absence of unacceptable toxicity.
  Disease subgroup: ALL Tumor Burden: high Dose level: 2 up to 2x106 EGFR+ cells/kg
  Autologous Anti-CD19CAR-4-1BB-CD3zeta-EGFRt-expressing T Lymphocytes: Given IV
- ALL (High Tumor Burden) Dose Level 3: Patients receive anti-CD19-CAR lentiviral vector-transduced autologous T cells IV over 20-30 minutes on day 0. Treatment may be repeated in no less than 21 days with or without additional lymphodepleting chemotherapy if there is persistent disease in the absence of unacceptable toxicity.
  Disease subgroup: ALL Tumor Burden: high Dose level: 3 up to 2x107 EGFR+ cells/kg
  Autologous Anti-CD19CAR-4-1BB-CD3zeta-EGFRt-expressing T Lymphocytes: Given IV
- ALL (Low Tumor Burden) Dose Level 1: Patients receive anti-CD19-CAR lentiviral vector-transduced autologous T cells IV over 20-30 minutes on day 0. Treatment may be repeated in no less than 21 days with or without additional lymphodepleting chemotherapy if there is persistent disease in the absence of unacceptable toxicity.
  Disease subgroup: ALL Tumor Burden: low Dose level: 1 up to 2x105 EGFR+ cells/kg
  Autologous Anti-CD19CAR-4-1BB-CD3zeta-EGFRt-expressing T Lymphocytes: Given IV
- CLL Dose Level 1: Patients receive anti-CD19-CAR lentiviral vector-transduced autologous T cells IV over 20-30 minutes on day 0. Treatment may be repeated in no less than 21 days with or without additional lymphodepleting chemotherapy if there is persistent disease in the absence of unacceptable toxicity.
  Disease subgroup: CLL Dose level: 1 up to 2x105 EGFR+ cells/kg
  Autologous Anti-CD19CAR-4-1BB-CD3zeta-EGFRt-expressing T Lymphocytes: Given IV
- CLL Dose Level 2: Patients receive anti-CD19-CAR lentiviral vector-transduced autologous T cells IV over 20-30 minutes on day 0. Treatment may be repeated in no less than 21 days with or without additional lymphodepleting chemotherapy if there is persistent disease in the absence of unacceptable toxicity.
  Disease subgroup: CLL Dose level: 2 up to 2x106 EGFR+ cells/kg
  Autologous Anti-CD19CAR-4-1BB-CD3zeta-EGFRt-expressing T Lymphocytes: Given IV
- CLL Dose Level 3: Patients receive anti-CD19-CAR lentiviral vector-transduced autologous T cells IV over 20-30 minutes on day 0. Treatment may be repeated in no less than 21 days with or without additional lymphodepleting chemotherapy if there is persistent disease in the absence of unacceptable toxicity.
  Disease subgroup: CLL Dose level: 3 up to 2x107 EGFR+ cells/kg
  Autologous Anti-CD19CAR-4-1BB-CD3zeta-EGFRt-expressing T Lymphocytes: Given IV
- CLL (Ibrutinib) Dose Level 2: Patients receive anti-CD19-CAR lentiviral vector-transduced autologous T cells IV over 20-30 minutes on day 0. Treatment may be repeated in no less than 21 days with or without additional lymphodepleting chemotherapy if there is persistent disease in the absence of unacceptable toxicity.
  Disease subgroup: CLL (ibrutinib) Dose level: 2 up to 2x106 EGFR+ cells/kg
  Autologous Anti-CD19CAR-4-1BB-CD3zeta-EGFRt-expressing T Lymphocytes: Given IV
- NHL Dose Level 1: Patients receive anti-CD19-CAR lentiviral vector-transduced autologous T cells IV over 20-30 minutes on day 0. Treatment may be repeated in no less than 21 days with or without additional lymphodepleting chemotherapy if there is persistent disease in the absence of unacceptable toxicity.
  Disease subgroup: NHL Dose level: 1 up to 2x105 EGFR+ cells/kg
  Autologous Anti-CD19CAR-4-1BB-CD3zeta-EGFRt-expressing T Lymphocytes: Given IV
- NHL Dose Level 2; NHL (Dose Dense) Dose Level 2: Patients receive anti-CD19-CAR lentiviral vector-transduced autologous T cells IV over 20-30 minutes on day 0. Treatment may be repeated in no less than 21 days with or without additional lymphodepleting chemotherapy if there is persistent disease in the absence of unacceptable toxicity.
  Disease subgroup: NHL Dose level: 2 up to 2x106 EGFR+ cells/kg
  Autologous Anti-CD19CAR-4-1BB-CD3zeta-EGFRt-expressing T Lymphocytes: Given IV
- NHL Dose Level 3: Patients receive anti-CD19-CAR lentiviral vector-transduced autologous T cells IV over 20-30 minutes on day 0. Treatment may be repeated in no less than 21 days with or without additional lymphodepleting chemotherapy if there is persistent disease in the absence of unacceptable toxicity.
  Disease subgroup: NHL Dose level: 3 up to 2x107 EGFR+ cells/kg
  Autologous Anti-CD19CAR-4-1BB-CD3zeta-EGFRt-expressing T Lymphocytes: Given IV
Period: Overall Study
Arm/Group | ALL (High Tumor Burden) Dose Level 1 | ALL (High Tumor Burden) Dose Level 2 | ALL (High Tumor Burden) Dose Level 3 | ALL (Low Tumor Burden) Dose Level 1 | ALL (Low Tumor Burden) Dose Level 2 | CLL Dose Level 1 | CLL Dose Level 2 | CLL Dose Level 3 | CLL (Ibrutinib) Dose Level 2 | NHL Dose Level 1 | NHL Dose Level 2 | NHL Dose Level 3 | NHL (Dose Dense) Dose Level 2
Started | 39 | 5 | 2 | 1 | 18 | 5 | 22 | 1 | 20 | 5 | 49 | 10 | 20
Completed | 9 | 2 | 1 | 0 | 11 | 4 | 10 | 0 | 9 | 2 | 17 | 4 | 7
Not Completed | 30 | 3 | 1 | 1 | 7 | 1 | 12 | 1 | 11 | 3 | 32 | 6 | 13
Not completed — Death | 27 | 3 | 1 | 1 | 5 | 1 | 11 | 1 | 11 | 3 | 32 | 6 | 13
Not completed — Lost to Follow-up | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Patient proceeded to new therapy | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ALL (High Tumor Burden) Dose Level 1 | ALL (High Tumor Burden) Dose Level 2 | ALL (High Tumor Burden) Dose Level 3 | ALL (Low Tumor Burden) Dose Level 1 | ALL (Low Tumor Burden) Dose Level 2 | CLL Dose Level 1 | CLL Dose Level 2 | CLL Dose Level 3 | CLL (Ibrutinib) Dose Level 2 | NHL Dose Level 1 | NHL Dose Level 2 | NHL Dose Level 3 | NHL (Dose Dense) Dose Level 2 | Total
Number analyzed (Participants) | 39 | 5 | 2 | 1 | 18 | 5 | 22 | 1 | 20 | 5 | 49 | 10 | 20 | 197
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 35 | 5 | 1 | 1 | 15 | 4 | 17 | 1 | 12 | 4 | 40 | 8 | 15 | 158
  >=65 years | 4 | 0 | 1 | 0 | 3 | 1 | 5 | 0 | 8 | 1 | 9 | 2 | 5 | 39
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 2 | 2 | 1 | 8 | 2 | 7 | 0 | 6 | 2 | 13 | 2 | 5 | 66
  Male | 23 | 3 | 0 | 0 | 10 | 3 | 15 | 1 | 14 | 3 | 36 | 8 | 15 | 131
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 1 | 0 | 0 | 4 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 14
  Not Hispanic or Latino | 33 | 4 | 2 | 1 | 14 | 5 | 20 | 1 | 20 | 5 | 47 | 10 | 20 | 182
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 7
  Asian | 4 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 3 | 12
  Black or African American | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 4
  White | 31 | 4 | 2 | 0 | 13 | 4 | 19 | 1 | 19 | 5 | 45 | 10 | 14 | 167
  Mexican or Mexican American | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 4
  White American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 39 | 5 | 2 | 1 | 18 | 5 | 22 | 1 | 20 | 5 | 49 | 10 | 20 | 197

OUTCOME MEASURES:

1. Primary Outcome: Death Within 8 Weeks of the Study Cell Infusion Thought to be Definitely or Probably Related to Chimeric Antigen Receptor (CAR) T Cell Therapy
Description: Death within 8 weeks of the study cell infusion thought to be definitely or probably related to CAR T cell therapy will be assessed.
Time Frame: Within 8 weeks of the study cell infusion
Measure: Count of Participants; unit: Participants
Arm/Group | ALL (High Tumor Burden) Dose Level 1 | ALL (High Tumor Burden) Dose Level 2 | ALL (High Tumor Burden) Dose Level 3 | ALL (Low Tumor Burden) Dose Level 1 | ALL (Low Tumor Burden) Dose Level 2 | CLL Dose Level 1 | CLL Dose Level 2 | CLL Dose Level 3 | CLL (Ibrutinib) Dose Level 2 | NHL Dose Level 1 | NHL Dose Level 2 | NHL Dose Level 3 | NHL (Dose Dense) Dose Level 2
Number analyzed (Participants) | 39 | 5 | 2 | 1 | 18 | 5 | 22 | 1 | 20 | 5 | 49 | 10 | 20
Participants | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0

2. Primary Outcome: Dose Limiting Toxicities
Description: Outcome will be reported as a count of participants that experienced a dose limiting toxicity on the study within 30 days post infusion.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | ALL (High Tumor Burden) Dose Level 1 | ALL (High Tumor Burden) Dose Level 2 | ALL (High Tumor Burden) Dose Level 3 | ALL (Low Tumor Burden) Dose Level 1 | ALL (Low Tumor Burden) Dose Level 2 | CLL Dose Level 1 | CLL Dose Level 2 | CLL Dose Level 3 | CLL (Ibrutinib) Dose Level 2 | NHL Dose Level 1 | NHL Dose Level 2 | NHL Dose Level 3 | NHL (Dose Dense) Dose Level 2
Number analyzed (Participants) | 39 | 5 | 2 | 1 | 18 | 5 | 22 | 1 | 20 | 5 | 49 | 10 | 20
Participants | 3 | 1 | 1 | 0 | 2 | 0 | 4 | 0 | 1 | 0 | 0 | 3 | 0

3. Primary Outcome: Objective Response Rate of Complete Response and Partial Response
Description: Outcome will be reported as the count of patients per arm that experienced a complete response/partial response.
  Complete response (CR): CR per Lugano criteria for nodal disease and minimal residual disease (MRD)-negative CR by flow cytometry for marrow disease.
  Partial response (PR): > 50% reduction of the sum of the products of the perpendicular diameters of marker lesions, no progression of any existing lesions, and no new lesions.
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | ALL (High Tumor Burden) Dose Level 1 | ALL (High Tumor Burden) Dose Level 2 | ALL (High Tumor Burden) Dose Level 3 | ALL (Low Tumor Burden) Dose Level 1 | ALL (Low Tumor Burden) Dose Level 2 | CLL Dose Level 1 | CLL Dose Level 2 | CLL Dose Level 3 | CLL (Ibrutinib) Dose Level 2 | NHL Dose Level 1 | NHL Dose Level 2 | NHL Dose Level 3 | NHL (Dose Dense) Dose Level 2
Number analyzed (Participants) | 39 | 5 | 2 | 1 | 18 | 5 | 22 | 1 | 20 | 5 | 49 | 10 | 20
Participants | 32 | 5 | 1 | 1 | 18 | 4 | 16 | 1 | 12 | 2 | 28 | 4 | 10

4. Primary Outcome: Overall Survival
Description: Outcome will be reported as a count of patients who survived up to 1 year post infusion.
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | ALL (High Tumor Burden) Dose Level 1 | ALL (High Tumor Burden) Dose Level 2 | ALL (High Tumor Burden) Dose Level 3 | ALL (Low Tumor Burden) Dose Level 1 | ALL (Low Tumor Burden) Dose Level 2 | CLL Dose Level 1 | CLL Dose Level 2 | CLL Dose Level 3 | CLL (Ibrutinib) Dose Level 2 | NHL Dose Level 1 | NHL Dose Level 2 | NHL Dose Level 3 | NHL (Dose Dense) Dose Level 2
Number analyzed (Participants) | 39 | 5 | 2 | 1 | 18 | 5 | 22 | 1 | 20 | 5 | 49 | 10 | 20
Participants | 12 | 2 | 1 | 0 | 13 | 4 | 13 | 0 | 9 | 2 | 20 | 4 | 7

5. Primary Outcome: Progression Free Survival
Description: Outcome will be reported as the count of patients per arm that survived and whose disease did not progress in the 1 year timeframe post infusion.
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | ALL (High Tumor Burden) Dose Level 1 | ALL (High Tumor Burden) Dose Level 2 | ALL (High Tumor Burden) Dose Level 3 | ALL (Low Tumor Burden) Dose Level 1 | ALL (Low Tumor Burden) Dose Level 2 | CLL Dose Level 1 | CLL Dose Level 2 | CLL Dose Level 3 | CLL (Ibrutinib) Dose Level 2 | NHL Dose Level 1 | NHL Dose Level 2 | NHL Dose Level 3 | NHL (Dose Dense) Dose Level 2
Number analyzed (Participants) | 39 | 5 | 2 | 1 | 18 | 5 | 22 | 1 | 20 | 5 | 49 | 10 | 20
Participants | 2 | 0 | 0 | 0 | 1 | 3 | 4 | 0 | 2 | 0 | 4 | 1 | 2

6. Secondary Outcome: Duration of Persistence of Adoptively Transferred CD19 Chimeric Antigen Receptor (CAR)-T Cells
Description: Duration of persistence of adoptively transferred CD19 chimeric antigen receptor (CAR)-T cells. Outcome will be reported for each of the 3 cohorts on the study. Outcome data is both count of patients alive after 1 year and count of patients with CAR-T cells detected at 1 year.
Time Frame: Up to day 365
Population: Cohorts for this outcome are combined into disease type. The first row is a count of participants that were alive at the 1 year post infusion point within these cohorts. The second row is a count of participants who had CAR-T cells present at the 1 year follow up. This count has a lower number analyzed because it is out of the participants who had available CAR-T data at the 1 year followup timepoint.
Measure: Count of Participants; unit: Participants
Groups:
- Acute Lymphocytic Leukemia Cohort: Cohort containing all ALL subtypes and treatment dose levels.
- Non-Hodgkin Lymphoma Cohort: Cohort containing all NHL subtypes and treatment dose levels.
- Chronic Lymphocytic Leukemia Cohort: Cohort containing all CLL subtypes and treatment dose levels.
Arm/Group | Acute Lymphocytic Leukemia Cohort | Non-Hodgkin Lymphoma Cohort | Chronic Lymphocytic Leukemia Cohort
Number analyzed (Participants) | 65 | 84 | 48
Participants
  Count of patients alive 1 year after CAR-T cell infusion | 33 | 46 | 23
  Count of patients with CAR-T cells detected at 1 year: number analyzed (Participants) | 29 | 34 | 22
  Count of patients with CAR-T cells detected at 1 year | 3 | 14 | 13

7. Secondary Outcome: Migration of Adoptively Transferred CD19 Chimeric Antigen Receptor (CAR)-T Cells
Description: Migration of adoptively transferred CD19 chimeric antigen receptor (CAR)-T cells. Outcome will be reported for each of the 3 cohorts on the study. Outcome data is both count of patients with bone marrow disease involvement and count of patients with CAR-T cells detected in bone marrow at restaging.
Time Frame: Up to 1 year
Population: This outcome is split into arms by disease type. The first row is a count of participants out of those treated that had bone marrow disease involvement. The second row reports the count of participants with CAR-T cells detected in bone marrow at restaging. The total number analyzed for the count of participants with CAR-T cells detected in bone marrow at restaging is lower than the overall number analyzed because it is those who had available bone marrow data at the time of restaging.
Measure: Count of Participants; unit: Participants
Arm/Group | Acute Lymphocytic Leukemia Cohort | Non-Hodgkin Lymphoma Cohort | Chronic Lymphocytic Leukemia Cohort
Number analyzed (Participants) | 65 | 84 | 48
Participants
  Count of patients with bone marrow disease involvement | 62 | 24 | 47
  Count of patients with CAR-T cells detected in bone marrow at restaging: number analyzed (Participants) | 51 | 19 | 40
  Count of patients with CAR-T cells detected in bone marrow at restaging | 49 | 15 | 37

ADVERSE EVENTS:
Time Frame: Adverse events will be assessed up to 1 year for each patient following their infusion.
Description: Adverse Events will be extracted from the patient record and assessed by the Principle Investigator for relation to treatment. AEs will beb graded in severity according to the NCI Common Terminology Criteria for Adverse Events (CTCAE v4.03).
Arm/Group | ALL (High Tumor Burden) Dose Level 1 | ALL (High Tumor Burden) Dose Level 2 | ALL (High Tumor Burden) Dose Level 3 | ALL (Low Tumor Burden) Dose Level 1 | ALL (Low Tumor Burden) Dose Level 2 | CLL Dose Level 1 | CLL Dose Level 2 | CLL Dose Level 3 | CLL (Ibrutinib) Dose Level 2 | NHL Dose Level 1 | NHL Dose Level 2 | NHL Dose Level 3 | NHL (Dose Dense) Dose Level 2
All-Cause Mortality (participants affected / at risk) | 27/39 | 3/5 | 1/2 | 1/1 | 5/18 | 1/5 | 11/22 | 1/1 | 11/20 | 3/5 | 32/49 | 6/10 | 13/20
Serious Adverse Events (participants affected / at risk) | 39/39 | 5/5 | 2/2 | 0/1 | 14/18 | 5/5 | 22/22 | 1/1 | 20/20 | 5/5 | 49/49 | 7/10 | 20/20
Other Adverse Events (participants affected / at risk) | 39/39 | 5/5 | 2/2 | 1/1 | 18/18 | 5/5 | 22/22 | 1/1 | 20/20 | 5/5 | 49/49 | 10/10 | 19/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALL (High Tumor Burden) Dose Level 1 (N=39) | ALL (High Tumor Burden) Dose Level 2 (N=5) | ALL (High Tumor Burden) Dose Level 3 (N=2) | ALL (Low Tumor Burden) Dose Level 1 (N=1) | ALL (Low Tumor Burden) Dose Level 2 (N=18) | CLL Dose Level 1 (N=5) | CLL Dose Level 2 (N=22) | CLL Dose Level 3 (N=1) | CLL (Ibrutinib) Dose Level 2 (N=20) | NHL Dose Level 1 (N=5) | NHL Dose Level 2 (N=49) | NHL Dose Level 3 (N=10) | NHL (Dose Dense) Dose Level 2 (N=20)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 30 (42) | 5 (5) | 2 (2) | 0 (0) | 10 (11) | 4 (5) | 21 (26) | 1 (1) | 10 (10) | 3 (3) | 27 (34) | 7 (10) | 12 (13)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Heart failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial tamponade (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sick sinus syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fever (General disorders) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Multi-organ failure (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sudden death NOS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 10 (10) | 5 (5) | 2 (2) | 0 (0) | 4 (4) | 1 (1) | 8 (8) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 5 (5) | 2 (2)
Anorectal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Central nervous system necrosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphasia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Edema cerebral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 2 (2)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Capillary leak syndrome (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 9 (9) | 5 (5) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 6 (6) | 5 (5) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALL (High Tumor Burden) Dose Level 1 (N=39) | ALL (High Tumor Burden) Dose Level 2 (N=5) | ALL (High Tumor Burden) Dose Level 3 (N=2) | ALL (Low Tumor Burden) Dose Level 1 (N=1) | ALL (Low Tumor Burden) Dose Level 2 (N=18) | CLL Dose Level 1 (N=5) | CLL Dose Level 2 (N=22) | CLL Dose Level 3 (N=1) | CLL (Ibrutinib) Dose Level 2 (N=20) | NHL Dose Level 1 (N=5) | NHL Dose Level 2 (N=49) | NHL Dose Level 3 (N=10) | NHL (Dose Dense) Dose Level 2 (N=20)
Anemia (Blood and lymphatic system disorders) | 33 (44) | 4 (4) | 1 (1) | 1 (2) | 12 (15) | 3 (6) | 19 (27) | 1 (1) | 16 (19) | 4 (6) | 32 (46) | 6 (7) | 14 (20)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 5 (6) | 4 (4) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 5 (5) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2)
Fatigue (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Fever (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localized edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anorectal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter related infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Lung infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreas infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 8 (8) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 4 (4) | 2 (2)
Alanine aminotransferase increased (Investigations) | 4 (4) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Alkaline phosphatase increased (Investigations) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 4 (4) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 5 (5) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 2 (2)
Cardiac troponin I increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
CPK increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT corrected interval prolonged (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Fibrinogen decreased (Investigations) | 6 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
GGT increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 39 (58) | 5 (5) | 2 (2) | 1 (2) | 18 (27) | 5 (7) | 21 (30) | 1 (1) | 20 (27) | 5 (8) | 48 (81) | 10 (14) | 19 (38)
Lymphocyte count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Neutrophil count decreased (Investigations) | 39 (59) | 5 (5) | 2 (2) | 1 (4) | 18 (25) | 5 (9) | 22 (34) | 1 (2) | 20 (29) | 5 (7) | 48 (68) | 10 (13) | 19 (31)
Platelet count decreased (Investigations) | 29 (52) | 5 (5) | 2 (2) | 1 (3) | 13 (17) | 5 (7) | 20 (28) | 1 (2) | 15 (17) | 4 (6) | 31 (43) | 5 (6) | 11 (18)
Urine output decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight gain (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 39 (56) | 5 (5) | 2 (2) | 1 (3) | 18 (24) | 5 (8) | 21 (31) | 1 (1) | 20 (29) | 5 (7) | 47 (67) | 10 (13) | 18 (28)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alkalosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 9 (12) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (2) | 4 (5) | 1 (1) | 4 (4) | 0 (0) | 4 (5) | 2 (2) | 4 (4)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2) | 4 (4) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 9 (9) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 5 (5) | 2 (2) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 7 (10) | 5 (5) | 1 (1) | 0 (0) | 9 (10) | 3 (4) | 11 (12) | 1 (1) | 4 (4) | 2 (2) | 21 (22) | 3 (4) | 7 (9)
Hypophosphatemia (Metabolism and nutrition disorders) | 15 (16) | 5 (5) | 2 (2) | 0 (0) | 6 (6) | 1 (1) | 10 (11) | 1 (1) | 5 (5) | 0 (0) | 14 (16) | 7 (8) | 5 (5)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Encephalopathy (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 4 (4) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Movements involuntary (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nystagmus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Personality change (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 3 (3) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 8 (8) | 1 (1) | 3 (3) | 0 (0) | 6 (7) | 2 (2) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Menopause (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 6 (6) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 5 (8) | 0 (0) | 7 (10) | 1 (1) | 8 (11) | 2 (2) | 4 (5)
Hypotension (Vascular disorders) | 12 (12) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 1 (2) | 6 (8) | 0 (0) | 9 (9) | 2 (2) | 8 (10) | 2 (3) | 3 (3)
Lymphedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2021-06-01): https://cdn.clinicaltrials.gov/large-docs/17/NCT01865617/Prot_000.pdf